CLINICAL TRIAL: NCT00049634
Title: A Phase I/II Study of Immunologically Engineered rhG-CSF Mobilized Peripheral Blood Stem Cells (PBSC) for Allogeneic Transplant From HLA Identical, Related Donors for Treatment of Myeloid Malignancies
Brief Title: Donor Peripheral Stem Cell Transplant in Treating Patients With Myelodysplastic Syndrome, Acute Myeloid Leukemia, or Myeloproliferative Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ann E. Woolfrey, Fred Hutchinson Cancer Research Center
Masking: None | Purpose: Treatment
Other Study IDs: 1628.00; FHCRC-1628.00; NCI-H02-0099; CDR0000258137 (Registry Identifier: PDQ)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; essential thrombocythemia; polycythemia vera; previously treated myelodysplastic syndromes; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Anemia, Refractory, with Excess of Blasts; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy drugs before a donor peripheral blood stem cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving colony-stimulating factors, such as G-CSF, to the donor helps the stem cells move from the bone marrow to the blood so they can be collected and stored.

PURPOSE: This phase I/II trial is studying how well donor peripheral stem cell transplant works in treating patients with myelodysplastic syndrome, acute myeloid leukemia, or myeloproliferative disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of grades II, III, and IV graft-vs-host disease (GVHD) in patients with myelodysplastic syndromes (MDS), acute myeloid leukemia transformed from MDS, or myeloproliferative disorders treated with immunologically engineered, filgrastim (G-CSF)-mobilized, allogeneic peripheral blood stem cell transplantation.
* Determine the incidence of graft failure, relapse, and transplant-related mortality by day 100 in patients treated with this regimen.
* Determine the incidence of chronic GVHD, in terms of number and duration of immunosuppressant therapies, in patients treated with this regimen.
* Determine the feasibility of partial T-cell depletion in G-CSF-mobilized peripheral blood stem cells.

OUTLINE: Patients receive conditioning with oral busulfan every 6 hours on days -7 to -4 and cyclophosphamide IV on days -3 and -2. Immunologically engineered, filgrastim (G-CSF)-mobilized, allogeneic peripheral blood stem cells are infused on day 0.

Patients receive graft-vs-host disease prophylaxis comprising methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV over 1-4 hours (orally twice daily when tolerated) on days -1 to 80 and then gradually tapered over 5 months beginning on day 81.

Patients are followed regularly through day 100 and then at 1 year.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Myelodysplastic syndromes (MDS) that has advanced beyond refractory anemia (RA)
  * RA with excess blasts (RAEB) (greater than 5% blasts)
  * RAEB in transformation (greater than 20% but less than 30% blasts)
  * Acute myeloid leukemia (greater than 30% blasts) that evolved from MDS
  * Myeloproliferative disorder, including chronic myelomonocytic leukemia, agnogenic myeloid metaplasia, polycythemia vera, or essential thrombosis
* No chronic myelogenous leukemia with or without excess (greater than 5%) blasts
* Must have an HLA-identical, related donor

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* Not specified

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin less than 2 times upper limit of normal (ULN)*
* SGOT/SGPT less than 2 times ULN* NOTE: * Unless due to malignancy

Renal

* Creatinine no greater than 2.0 mg/dL OR
* Glomerular filtration rate at least 60 mL/min

Cardiovascular

* Cardiac ejection fraction at least 45%

Pulmonary

* DLCO at least 60% of predicted

Other

* HIV negative
* Human antimouse antibody negative
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other medical condition that would preclude study participation
* No hypersensitivity to cyclosporine

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior marrow transplantation
* No concurrent growth factors for 21 days after study transplantation

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-01; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Incidence of grade II, III, and IV graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Woolfrey, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington